CLINICAL TRIAL: NCT06266819
Title: The Effect of Mint Flavored Chewing Gum Application on Nausea Vomiting Severity, Coping With Stress and Anxiety Level in Pregnants With Hyperemesis Gravidarum
Brief Title: The Effect of Mint Flavored Chewing Gum on Hyperemesis Gravidarum Nausea Vomiting Severity, Coping With Stress and Anxiety Level in Pregnants With Hyperemesis Gravidarum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Leyla Emirik, PhD Student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OU-HEM-LE-01
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hyperemesis Gravidarum
Keywords: hyperemesis gravidarum; chewing gum; nausea and vomiting; mint
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: two groups with chewing mint gum experimental group and a control group
Who Masked: Outcomes Assessor
Masking Description: The study protocol in the research will be created using SPIRIT as a guide. Reporting of the trial will be structured according to the CONSORT checklist. Random distribution of pregnant women included in the study to the intervention and control groups will be made at www.randomizer.org. Which group will be the intervention or control group will be determined by drawing lots at the beginning of the study. Pregnant women in the intervention group will be given the practice of chewing mint-flavored gum.
  Since the researcher knows which group the pregnant women are included in, the data collection phase of the study is single blind. To avoid selection bias in this study, pregnant women will be randomly assigned to the intervention and control groups by randomization method. To prevent reporting bias, the analysis of the research data will be carried out by an expert statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the chewing of a mint-flavored gum group (Experimental): In data collection, pregnant women will sign an informed consent form before the application. Personal Information Form, VAS Scale, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale will be filled out. In addition to the routine treatment plan, the application will begin at least 4 hours after the antiemetic administration. The application will continue by chewing mint-flavored gum twice a day for at least 15 minutes for 3 days. The VAS scale will be filled after the morning chewing application, and the VAS Scale, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale will be filled in after the evening application. The forms of patients discharged during this period will be filled in via phone.
  Interventions: Other: chewing gum
- control group (No Intervention): In data collection, pregnant women will sign an informed consent form before the application. At least 4 hours after the antiemetic administration, the Personal Information Form, VAS Scale, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale will be filled out. Routine treatment and nursing care will be applied to the control group, and no intervention will be performed. 1. After the forms are applied, the forms will continue to be filled for 3 days: VAS Scale in the morning, VAS Scale in the evening, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale. The forms of discharged patients will be filled in via phone.

INTERVENTIONS:
Other: chewing gum — In addition to the routine treatment plan, mint-flavored gum will be chewed for an average of 15 minutes at least 4 hours after the antiemetic application.
  Arms: the chewing of a mint-flavored gum group

SUMMARY:
In the research planned as a randomized controlled study, the experimental groups will be administered routine hyperemesis gravidarum (HG) treatment as well as chewing mint-flavored gum, while the control group will only receive routine HG treatment and no intervention will be performed. This study aims to contribute to the literature by investigating the effect of chewing mint-flavored gum on the severity of nausea and vomiting, coping with stress, and anxiety levels due to hyperemesis gravidarum in pregnant women.

DETAILED DESCRIPTION:
The data of the research will be collected after the necessary institutional permission and ethics committee approval have been obtained. Women who meet the inclusion criteria for the study will be informed about the method to be followed in the research. Those who want to participate in the research will read and sign the volunteer information form.

1. Intervention Group In data collection, pregnant women will sign an informed consent form before the application. Personal Information Form, VAS Scale, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale will be filled out. In addition to the routine treatment plan, the application will begin at least 4 hours after the antiemetic application (Gökbulut, 2021). The application will continue by chewing mint-flavored gum twice a day for at least 15 minutes for 3 days. The VAS scale will be filled after the morning chewing application, and the VAS Scale, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale will be filled in after the evening application. The forms of patients discharged during this period will be filled in via phone.
2. Control Group In data collection, pregnant women will sign an informed consent form before the application. At least 4 hours after the antiemetic application (Gökbulut, 2021), the Personal Information Form, VAS Scale, PUQE Scale and Stress Coping Styles Scale and State Anxiety Scale will be filled out. Routine treatment and nursing care will be applied to the control group, and no intervention will be performed. 1. After the forms are applied, the forms will continue to be filled for 3 days: VAS Scale in the morning, VAS Scale in the evening, PUQE Scale, Stress Coping Styles Scale and State Anxiety Scale. The forms of discharged patients will be filled in via phone.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and over
* At least primary school graduate
* The one who is married
* Pregnant women who are younger than 16 weeks of gestation and diagnosed with hyperemesis
* Those who agreed to participate in the study

Exclusion Criteria:

* Those with a history of chronic disease
* Having a health problem that may cause nausea and vomiting in the current pregnancy
* Those who are allergic to mint

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-Specific Nausea and Vomiting Severity Scale (PUQE-24) | 8 hours
  It was developed to evaluate the severity of pregnancy-specific nausea and vomiting in the last 24 hours. Pregnancy-Specific Nausea and Vomiting Severity Scale (PUQE-24) consists of 3 questions: "duration of nausea or stomach discomfort", "number of vomiting" and "number of retching". Answers to the questions are scored between 1-5 points. The total score of the scale is obtained by the sum of the scores of the answers given to the questions. The lowest score that can be obtained from the scale is 3 and the highest score is 15. If the total score obtained as a result of the PUQE-24 scoring system is 3-6, it is considered mild, 7-12 is considered moderate, and 13-15 is considered severe nausea and vomiting. The scale has no subdimensions. Cronbach's alpha value of the Turkish version of the scale is 0.75.
Visual Analog Scale (VAS) | 8 hours
  It is used for pain assessment in musculoskeletal and other clinical evaluations. VAS is used to convert some values that cannot be measured numerically into numerical values. It is a frequently used measurement tool because it is easy to apply and safe. At the left end of the 10 cm long horizontal line are the words 'I have no pain' and at the right end the words 'I have pain'. The individual is told to mark the point on this horizontal line that best expresses the intensity of pain in his body. The distance of the point marked by the individual to the left end is measured and the pain score is determined. As the VAS value approaches 10, the intensity of the pain increases, and as it approaches 0, the intensity decreases. The lowest score from the scale is 0 and the highest score is 10.

SECONDARY OUTCOMES:
Stress Coping Styles Scale (SCSS) | 8 hours
  Coping with Stress Coping Styles Scale is a four-point Likert type, consisting of 30 items and 5 subscales. Effective coping styles with stress are evaluated with the "Self-Confident Approach", "Optimistic Approach" and "Social Support Seeking Approach" sub-dimensions, while ineffective coping styles in coping with stress are evaluated with the "Helpless Approach" and "Submissive Approach" sub-dimensions. Higher scores indicate that the person uses more stress coping style. Cronbach Alpha Coefficients of the scale were found to be 0.78 for "Optimistic Approach", 0.83 for "Self-Security Approach", 0.90 for "Helpless Approach", 0.89 for "Submissive Approach" and 0.61 for "Seeking Social Support".
State-Trait Anxiety Inventory (STAI) | 8 hours
  State-Trait Anxiety Inventory (STAI) determines how an individual feels at a certain moment and condition. STAI consists of 20 items and answers are answered according to the degree of intensity of emotions or behaviors as (1) not at all, (2) a little, (3) a lot, (4) completely. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 in the scale are reverse scored. The STAI score is calculated by adding 50 points to the difference between the total weighted scores of direct statements and reverse statements. Scores between 20 and 80 can be obtained from STAI. If the score is below 36, it is considered that there is no anxiety, between 37 and 42 points, there is mild anxiety, and those with a score of 42 and above are considered to have high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Özel Şar Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No